CLINICAL TRIAL: NCT04980495
Title: A Phase 3b, Randomized, Open-label, Parallel-Group Study to Evaluate Different Dosing Regimens of Intravenous Efgartigimod to Maximize and Maintain Clinical Benefit in Patients With Generalized Myasthenia Gravis
Brief Title: An Open-label Study to Investigate the Clinical Efficacy of Different Dosing Regimens of Efgartigimod IV in Patients With Generalized Myasthenia Gravis
Acronym: ADAPT NXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2003; 2024-510932-36-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Generalized Myasthenia Gravis; MG - Myasthenia Gravis; gMG
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod IV - continuous regimen (Experimental): Participants receiving efgartigimod IV on a continuous regimen
  Interventions: Biological: Efgartigimod IV
- Efgartigimod IV - cyclic regimen (Experimental): Participants receiving efgartigimod IV on a cyclic regimen
  Interventions: Biological: Efgartigimod IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusions of efgartigimod

SUMMARY:
The purpose of this open-label study is to investigate the efficacy, safety, and tolerability of a continuous regimen of efgartigimod compared with a cyclic regimen in participants with Generalized Myasthenia Gravis (gMG).

Participants will receive efgartigimod throughout the study. The participants will be randomized to the continuous regimen arm or to the cyclic regimen arm. The study consists of a part A (regimen comparison period) where participants will continue the treatment based on the treatment regimen arm they were assigned at randomization. Following part A, participants will enter part B (extension period) where all participants will receive efgartigimod in the continuous regimen. The study duration for participants is up to 138 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, at the time of signing the informed consent.
* Diagnosed with Generalized Myasthenia Gravis (gMG) with confirmed documentation and supported by a physical exam and confirmed seropositivity for anti-acetylcholine receptor antibodies (AChR-Abs).
* Meets the clinical criteria as defined by the Myasthenia Gravis Foundation of America (MGFA) class II, III, or IV

Exclusion Criteria:

* Any other condition that, in the opinion of the investigator, would interfere with an accurate assessment of the clinical symptoms of gMG and/or put the participant at undue risk
* A thymectomy within 3 months of screening
* Use of the following prior or concomitant therapies:

  1. intravenous immunoglobulin (IVIg) or subcutaneous immunoglobulin (SCIg) within 14 days of day 1
  2. Rituximab within 6 months of day 1
  3. Eculizumab within 1 month of day 1
  4. Other monoclonal antibodies (eg, adalimumab, tocilizumab, ixekizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Mean of the average MG-ADL total score change from baseline during the visit of week 1 through week 21 by regimen arm | Up to 21 weeks
  The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The total score varies between 0 and 24, with higher total scores indicating more impairment.

SECONDARY OUTCOMES:
Incidence of AEs, SAEs and AESIs | Up to 136 weeks
  AE : adverse event; SAE: serious adverse event; AESI: adverse event of special interest
Change from baseline in the MG-ADL total score over time | Up to 126 weeks
  The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The total score varies between 0 and 24, with higher total scores indicating more impairment.
Normalized area under the effect curve (AUEC) of MG-ADL total score improvement from baseline | Up to 21 weeks
  The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The total score varies between 0 and 24, with higher total scores indicating more impairment.
Characterization of MG-ADL total score change from baseline | Up to 21 weeks
  The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The total score varies between 0 and 24, with higher total scores indicating more impairment.
Percentage of participants who have a ≥ 2, 3, 4, or 5 points improvement in MG-ADL total score from baseline | Up to 21 weeks
  The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The total score varies between 0 and 24, with higher total scores indicating more impairment.
Percentage of time participants have a change in MG-ADL total score of at least 2 points from baseline during Week 4 through Week 21 | Up to 21 weeks
  The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The total score varies between 0 and 24, with higher total scores indicating more impairment.
Percentage of participants who achieve MSE, defined as a MG-ADL total score of 0 or 1 | Up to 21 weeks
  MSE = minimal symptom expression; The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The total score varies between 0 and 24, with higher total scores indicating more impairment.

CONTACTS AND LOCATIONS:
Locations (39):
- United States (12):
  - Investigator Site 10 - US0010007, Carlsbad, California
  - Investigator Site 7 - US0010001, Orange, California
  - Investigator Site 9 - 0010006, Boca Raton, Florida
  - Investigator Site 15 - US0010014, Coral Springs, Florida
  - Investigator Site 16 - US0010009, Augusta, Georgia
  - Investigator Site 8 - US0010003, Chicago, Illinois
  - Investigator Site 6 - US0010008, Meadows, Illinois
  - Investigator Site 12 - US0010004, Kansas City, Kansas
  - Investigator Site 13 - US0010013, Portland, Oregon
  - Investigator Site 17 - US0010012, Philadelphia, Pennsylvania
  - Investigator Site 11 - US0010011, Austin, Texas
  - Investigator Site 14 - US0010010, Richmond, Virginia
- Austria (2):
  - Investigator Site 26 - AT0430002, Innsbruck
  - Investigator Site 27 - AT0430001, Vienna
- Investigator Site 28 - BE0320001, Leuven, Belgium
- Canada (2):
  - Investigator Site 29 - CA0019003, London
  - Investigator site 37 - CA0019002, Québec
- France (5):
  - Investigator Site 23 - FR0330005, Bordeaux
  - Investigator Site 24 - FR0330004, Lille
  - Investigator Site 20 - FR0330001, Marseille
  - Investigator Site 25 - FR0330003, Nice
  - Investigator site 38 - FR0330002, Paris
- Georgia (3):
  - Investigator Site 2 - GEO9950002, Tbilisi
  - Investigator Site 1 - GEO9950001, Tbilisi
  - Investigator Site 3 - GEO9950003, Tbilisi
- Germany (4):
  - Investigator Site 33 - DE0490004, Berlin
  - Investigator Site 36 - DE0490002, Bochum
  - Investigator Site 32 - DE0490001, Essen
  - Investigator Site 34 - DE0490005, Hanover
- Italy (5):
  - Investigator Site 31 - IT0390005, Bologna
  - Investigator Site 30 - IT0390004, Genova
  - Investigator Site 21 - IT0390002, Milan
  - Investigator site 39 - IT0390006, Pisa
  - Investigator Site 22 - IT0390001, Roma
- Investigator Site 35 - NL0310001, Amsterdam, Netherlands
- Poland (2):
  - Investigator Site 5 - PL0480002, Krakow
  - Investigator Site 4 - PL0480001, Lubin
- Spain (2):
  - Investigator Site 18 - ES0340002, Santiago de Compostela, A Coruña
  - Investigator Site 19 - ES0340001, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided